CLINICAL TRIAL: NCT06101173
Title: A Randomized, Observer-Blind, Positive-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Trivalent Poliomyelitis Vaccine (Sf-RVN Cell) in Healthy Adults Aged 18-54 Years
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Recombinant Trivalent Poliomyelitis Vaccine (Sf-RVN Cell) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-VLP-001
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Poliomyelitis
Keywords: Vaccine; Trivalent; Immunogenicity; Safety; ≥18 years
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental vaccine group A, Low dose, Intramuscular injection (IM) (Experimental): 1 dose of Low-adjuvant dose VLP-Polio vaccine on Visit 1
  Interventions: Biological: Recombinant Trivalent Poliomyelitis Vaccine (Sf-RVN Cell) (VLP-Polio)
- Control vaccine group A, IM (Active Comparator): 1 dose of IPOL vaccine on Visit 1
  Interventions: Biological: Inactivated poliomyelitis vaccine (IPOL)
- Experimental vaccine group B, Medium dose, Intramuscular injection (IM) (Experimental): 1 dose of Medium dose VLP-Polio vaccine on Visit 1
  Interventions: Biological: VLP-Polio
- Control vaccine group B, IM (Active Comparator): 1 dose of IPOL vaccine on Visit 1
  Interventions: Biological: IPOL
- Experimental vaccine group C, High dose, Intramuscular injection (IM) (Experimental): 1 dose of High dose VLP-Polio vaccine on Visit 1
  Interventions: Biological: VLP-Polio
- Control vaccine group C, IM (Active Comparator): 1 dose of IPOL vaccine on Visit 1
  Interventions: Biological: IPOL

INTERVENTIONS:
Biological: Recombinant Trivalent Poliomyelitis Vaccine (Sf-RVN Cell) (VLP-Polio) — 1 dose of VLP-Polio vaccine (0.5ml) on Visit 1
  Arms: Experimental vaccine group A, Low dose, Intramuscular injection (IM)
Biological: Inactivated poliomyelitis vaccine (IPOL) — 1 dose of IPOL vaccine (0.5ml) on Visit 1
  Arms: Control vaccine group A, IM
Biological: VLP-Polio — 1 dose of VLP-Polio vaccine (0.5ml) on Visit 1
  Arms: Experimental vaccine group B, Medium dose, Intramuscular injection (IM)
Biological: IPOL — 1 dose of IPOL vaccine (0.5ml) on Visit 1
  Arms: Control vaccine group B, IM
Biological: VLP-Polio — 1 dose of VLP-Polio vaccine (0.5ml) on Visit 1
  Arms: Experimental vaccine group C, High dose, Intramuscular injection (IM)
Biological: IPOL — 1 dose of IPOL vaccine (0.5ml) on Visit 1
  Arms: Control vaccine group C, IM

SUMMARY:
This is a randomized, observer-blind, positive-controlled study. There will be 3 treatment groups, in each treatment group, participants will be randomly assigned to receive either investigational vaccine (Low-adjuvant dose VLP-Polio, Medium dose VLP-Polio, or High dose VLP-Polio that are defined as Dose A, Dose M, and Dose H, respectively) or control vaccine in a ratio of 3:1 in each group. Distribution of participant's gender should be balanced in each group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers aged 18 to 54 years at time of screening.
* Participants who can understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent.
* Healthy or in stable health participants with pre-existing, stable, well-controlled disease, defined as mild disease or medical condition not requiring medical therapy or not requiring a change in medical therapy due to worsening of disease during the 6 months before enrollment may be enrolled at the discretion of the investigator.
* Female participants of childbearing potential must have a negative pregnancy test at screening and before the administration of investigational vaccine and have been using/ agree to use an adequate form of contraception 30 days prior to screening until 180 days post administration.
* Male participants must agree to use adequate contraception 30 days prior to screening until 180 days after the vaccination.

Exclusion Criteria:

* Tympanic temperature >37.4°C.
* Evidence of excessive alcohol or drug abuse.
* Have received any polio vaccines within 6 months prior to screening.
* History of severe allergic reaction (e.g., anaphylaxis) to any component of the vaccine.
* Pregnant or lactating at screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
* History of epilepsy or convulsions.
* Have developmental cognitive disability, dementia, or intellectual disabilities.
* Immune deficiency or immune suppressive treatment or auto-immune disease. For corticosteroids, a prednisone dose of <20 mg/day or equivalent is allowed. Inhaled and topical corticosteroids are allowed.
* Current diagnosis of polio or history of polio infection.
* Positive for HIV, Hepatitis B or Hepatitis C.
* Positive for COVID-19 test.
* Bleeding disorders or the usage of anticoagulants.
* Have received any other immunizations within 14 days prior to screening.
* Suffering from serious chronic disease or the disease is in progress and cannot be controlled, such as thyroid diseases (excluding thyroid nodules).
* Have received blood products within the past 3 months or plan to receive during the study period.
* Participate in other studies within 30 days (<30 days) before and/or during the study period.
* Abnormal safety laboratory parameters during the screening window that are clinically significant as per the judgement of the investigator.
* Any other factors that might interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participants to participate, in the opinion of the treating investigator.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited adverse reactions (AEs) within 7 days post vaccination. | Within 7 days post vaccination

SECONDARY OUTCOMES:
Occurrence of unsolicited AEs within 28 days post-vaccination. | Within 28 days post-vaccination
Occurrence of solicited AEs within 30 mins post-vaccination. | Within 30 mins post-vaccination
Occurrence of abnormal safety laboratory parameters on Day 3, Day 8. | Day 3, Day 8 post-vaccination
Occurrence of serious adverse events (SAEs) during the study period. | Through study completion, an average of 6 months
Geometric mean titer (GMT) of neutralizing antibodies against poliovirus type 1, 2, and 3 on Day 1 before vaccination and Day 29 and Day 180 after the vaccination. | Day 1 before vaccination and Day 29 and Day 180 after the vaccination
Geometric mean fold increase (GMI) of neutralizing antibodies against poliovirus type 1, 2, and 3 on Day 1 before vaccination and Day 29 and Day 180 after the vaccination. | Day 1 before vaccination and Day 29 and Day 180 after the vaccination
Seroconversion rate of neutralizing antibodies against poliovirus type 1, 2, and 3 on Day 1 before vaccination and Day 29 and Day 180 after the vaccination. | Day 1 before vaccination and Day 29 and Day 180 after the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chang, Dr, Principal Investigator — Nucleus Network Pty Ltd.
Locations (2):
- Australia (2):
  - Nucleus Network Pty Ltd, Geelong, Victoria
  - Nucleus Network Pty Ltd, Melbourne, Victoria